CLINICAL TRIAL: NCT02960230
Title: H3.3K27M Specific Peptide Vaccine Combined With Poly-ICLC With and Without PD-1 Inhibition Using Nivolumab for the Treatment of Newly Diagnosed HLA-A2 (02:01)+ H3.3K27M Positive Diffuse Intrinsic Pontine Glioma (DIPG) and Newly Diagnosed HLA-A2 (02:01)+ H3.3K27M Positive Gliomas
Brief Title: H3.3K27M Peptide Vaccine With Nivolumab for Children With Newly Diagnosed DIPG and Other Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sabine Mueller, MD, PhD (Other)
Collaborators: The V Foundation for Cancer Research (Other); Pacific Pediatric Neuro-Oncology Consortium (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Sabine Mueller, MD, PhD, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNOC 007; 150819 (Other: University of California, San Francisco); NCI-2017-01830 (Other: Clinical Trials Reporting Program (CTRP)); CA209-8TX (Other: Bristol-Meyers Squibb)
Record Dates: First submitted 2016-11-02; First posted 2016-11-09 (Estimated); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Glioma; Diffuse Midline Glioma, H3 K27M-Mutant
Keywords: peptide vaccine; immunotherapy; DIPG; vaccine; nivolumab
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Glioma | interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Stratum A: Newly Diagnosed DIPG (Experimental): Newly diagnosed children with diffuse intrinsic pontine glioma who are positive for HLA-A2 and the H3.3K27M mutation that underwent radiation therapy will receive the specific H3.3K27M peptide vaccine, combined with the tetanus toxoid (TT) peptide, emulsified in Montanide. Poly-ICLC, which is a synthetic nucleic acid, will be given concurrently to improve the therapeutic effects of the vaccine. Vaccine will be given every 3 weeks for the first 24 weeks, then if there is stable or improved disease, will be given every 6 weeks for a total treatment period of 96 weeks.
  Interventions: Biological: K27M peptide
- Stratum B: Newly Diagnosed Glioma (non-DIPG) (Experimental): Newly diagnosed children with gliomas other than DIPG who are positive for HLA-A2 and the H3.3K27M mutation that underwent radiation therapy will receive the specific H3.3K27M peptide vaccine, combined with the tetanus toxoid peptide, emulsified in Montanide. Poly-ICLC, which is a synthetic nucleic acid, will be given concurrently to improve the therapeutic effects of the vaccine. Vaccine will be given every 3 weeks for the first 24 weeks, then if there is stable or improved disease, will be given every 6 weeks for a total treatment period of 96 weeks.
  Interventions: Biological: K27M peptide
- Stratum C: Newly Diagnosed DIPG or other Midline Glioma (Experimental): Newly diagnosed children with DIPG or other midline gliomas (excluding primary spinal cord tumors) who are positive for HLA-A2 (02:01) and the H3.3K27M mutation that underwent radiation therapy will receive the specific H3.3K27M peptide vaccine, combined with the tetanus toxoid peptide, emulsified in Montanide. Poly-ICLC, which is a synthetic nucleic acid, will be given concurrently to improve the therapeutic effects of the vaccine. Nivolumab will also be given via IV. Vaccine will be given every 3 weeks for the first 24 weeks, then if there is stable or improved disease, will be given every 6 weeks for a total treatment period of 96 weeks. Nivolumab will continue to be given every 3 weeks throughout all of treatment.
  Interventions: Biological: K27M peptide; Drug: Nivolumab

INTERVENTIONS:
Biological: K27M peptide — K27M peptide vaccine, combined with Tetanus Toxoid peptide, emulsified in montanide. Poly-ICLC will be given concurrently
Drug: Nivolumab — anti-programmed cell death protein 1 (PD-1) monoclonal antibody
  Other Names: Keytruda
  Arms: Stratum C: Newly Diagnosed DIPG or other Midline Glioma

SUMMARY:
This is 3-arm, multicenter study that will be conducted through the Pacific Pediatric Neuro-oncology Consortium (PNOC). This study will assess the safety and immune activity of a synthetic peptide vaccine specific for the Histone 3 lysine27-to-methionine (H3.3K27M) epitope given in combination with poly-ICLC and the H3.3K27M epitope given in combination with poly-ICLC and the PD-1 inhibitor, nivolumab, in HLA-A2 (02:01)+ children with newly diagnosed diffuse intrinsic pontine glioma (DIPG) or other midline gliomas that are positive for H3.3K27M.

DETAILED DESCRIPTION:
Participants who are eligible will receive a specific peptide vaccine, along with a helper drug called poly-ICLC, in combination with nivolumab, every 3 weeks for the first 6 months of treatment. Participants will be monitored routinely by laboratory assessments, physical evaluation, vital signs, and MRI. Participants who tolerate therapy well and have stable or improved disease after 6 months of treatment can continue to receive treatment, nivolumab continuing every 3 weeks but vaccine and poly-ICLC now every 6 weeks, for a total of 96 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stratum A:

  • Newly diagnosed children (3-21 years old) with DIPG who are positive for the H3.3K27M mutation (positive testing in Clinical Laboratory Improvement Amendments (CLIA) laboratory) that underwent standard radiation therapy.
* Stratum B:

  • Newly diagnosed children (3-21 years old) with diagnosis of glioma other than DIPG who are positive for the H3.3K27M mutation (positive testing in CLIA laboratory) including spinal cord gliomas that underwent standard radiation therapy.
* Stratum C:

  * Newly diagnosed children 3-21 years of age with diagnosis of DIPG or midline glioma other than DIPG (excluding primary spinal cord gliomas) who are positive for the H3.3K27M mutation (positive testing from a CLIA or equivalent laboratory required), that underwent standard radiation therapy.

The following eligibility criteria apply to strata A, B and C:

* The patient must test positive for HLA-A*02:01 (positive testing from a CLIA or equivalent laboratory required; only the HLA A*02:01 subtype is eligible; other subtypes are excluded)
* The patient must be either off systemic steroids or be on stable dose of dexamethasone or equivalent (max 0.1 mg/kg/day; maximum 4mg/day) at time of enrollment.
* Patients must not have received any prior chemotherapy, immunotherapy or bone marrow transplant for the treatment of their tumor. Prior use of temozolomide during radiation at maximum of the standard pediatric dosing (defined as 90 mg/m^2/dose continuously during radiation therapy for 42 days) or dexamethasone is allowed.
* Patients must have undergone radiation therapy and surgery as part of their standard of care.

  * Stratum A: Radiation therapy must have started within 4 weeks of diagnosis by imaging or surgery, whichever is later.
  * Stratum B: For subjects undergoing surgery for more extensive resection, radiation therapy should be started within 4-6 weeks from surgery.
  * Stratum C: Radiation therapy must have started within 4 weeks of diagnosis by imaging or surgery, whichever is later. For subjects undergoing surgery for more extensive resection, radiation therapy should be started within 4-6 weeks from surgery.
* Karnofsky ≥ 50 for patients ≥ 16 years of age, and Lansky ≥ 50 for patients < 16 years of age (See Appendix A). Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* The patient must have adequate organ function defined as

Adequate Bone Marrow Function Defined as:

* Peripheral absolute neutrophil count (ANC) ≥ 1000/mm3 and
* Platelet count ≥ 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).

Adequate Renal Function Defined as:

* Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70 mL/min/1.73 m2 or
* A serum creatinine based on age/gender as follows:

Age Maximum Serum Creatinine (mg/dL) Male Female 3 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4 The threshold creatinine values in this table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the Center for Disease Control (CDC).

Adequate Liver Function Defined as:

* Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age and
* serum glutamic-pyruvic transaminase (SGPT)/ alanine aminotransferase (ALT) ≤ 110 U/L and
* Serum albumin ≥ 2 g/dL.

Adequate Pancreatic Function Defined as:

• Serum lipase ≤ ULN at baseline.

Adequate Pulmonary Function Defined as:

• No evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficiency, and a pulse oximetry of > 92% while breathing room air.

Adequate Neurologic Function Defined as:

* Patients with seizure disorder may be enrolled if seizure disorder is well controlled.
* The effects of the H3.3K27M vaccine and nivolumab on the developing human fetus are unknown. For this reason, females of child-bearing potential and males must agree to use adequate contraception. Adequate methods include: hormonal or barrier method of birth control; or abstinence prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Males treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for the duration of study participation.
* Ability to understand a written informed consent document, and the willingness to sign it. Assent will be obtained when appropriate based on the subjects age.

Exclusion Criteria:

* Investigational Drugs

  * Patients who are currently receiving another investigational drug are not eligible.
  * Prior treatment with another investigational drug.
* Anti-cancer Agents

  * Patients who are currently receiving other anti-cancer agents are not eligible.
  * Prior treatment with other anti-cancer agents.
* Patients who have received a live / attenuated vaccine within 30 days of first treatment.
* Patients with evidence of disseminated or leptomeningeal disease.
* Patients with a known disorder that affects their immune system, such as HIV or Hepatitis B or C, or an auto-immune disorder requiring systemic cytotoxic or immunosuppressive therapy are not eligible. Note: Patients that are currently using inhaled, intranasal, ocular, topical or other non-oral or non-IV steroids are not necessarily excluded from the study but need to be discussed with the study chair.
* Patients with a ≥ Grade 2 hypothyroidism due to history of autoimmunity are not eligible. (Note: Hypothyroidism due to previous irradiation or thyroidectomy will not impact eligibility).
* Patients who have received prior solid organ or bone marrow transplantation are not eligible.
* Patients with uncontrolled infection.
* Female patients of childbearing potential must not be pregnant or breast-feeding. Female patients of childbearing potential must have a negative serum or urine pregnancy test prior to the start of therapy (as clinically indicated).

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, MAS, Study Chair — University of California, San Francisco; Hideho Okada, MD, PhD, Study Chair — University of California, San Francisco
Locations (15):
- United States (14):
  - Rady Children's Hospital-San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- The University Children's Hospital in Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mueller S, Taitt JM, Villanueva-Meyer JE, Bonner ER, Nejo T, Lulla RR, Goldman S, Banerjee A, Chi SN, Whipple NS, Crawford JR, Gauvain K, Nazemi KJ, Watchmaker PB, Almeida ND, Okada K, Salazar AM, Gilbert RD, Nazarian J, Molinaro AM, Butterfield LH, Prados MD, Okada H. Mass cytometry detects H3.3K27M-specific vaccine responses in diffuse midline glioma. J Clin Invest. 2020 Dec 1;130(12):6325-6337. doi: 10.1172/JCI140378. PMID 32817593

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum A: Newly Diagnosed DIPG: Newly diagnosed children with diffuse intrinsic pontine glioma (DIPG) who are positive for HLA-A2 and the H3.3.K27M mutation that underwent radiation therapy will receive the specific H3.3.K27M peptide vaccine, combined with the tetanus toxoid (TT) peptide, emulsified in Montanide. Poly-ICLC, which is a synthetic nucleic acid, will be given concurrently to improve the therapeutic effects of the vaccine. Vaccine will be given every 3 weeks for the first 24 weeks, then if there is stable or improved disease, will be given every 6 weeks for a total treatment period of 96 weeks.
Period: Overall Study
Arm/Group | Stratum A: Newly Diagnosed DIPG | Stratum B: Newly Diagnosed Glioma (Non-DIPG) | Stratum C: Newly Diagnosed DIPG or Other Midline Glioma
Started | 19 | 10 | 21
Completed | 19 | 10 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum A: Newly Diagnosed DIPG | Stratum B: Newly Diagnosed Glioma (Non-DIPG) | Stratum C: Newly Diagnosed DIPG or Other Midline Glioma | Total
Number analyzed (Participants) | 19 | 10 | 21 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.11 (3.09) | 12.0 (3.62) | 9.38 (3.53) | 10.18 (3.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 10 | 26
  Male | 9 | 4 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 2 | 14
  Not Hispanic or Latino | 12 | 0 | 16 | 28
  Unknown or Not Reported | 4 | 1 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 10 | 7 | 18 | 35
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 7 | 1 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 19 | 10 | 15 | 44
  Switzerland | 0 | 0 | 6 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AE) Related to Treatment
Description: Safety of the vaccine (Strata A and B) or vaccine in combination with nivolumab (Stratum C) will be assessed for participants who received the vaccination. The severity of toxicities will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE)version 5.0. and include any clinically-significant lab abnormalities meeting Grade 3, 4, or 5 criteria according to CTCAE. Grade 1 & 2 AEs will be summarized if probably, possible, or definitely related to study therapy. Descriptive statistics will be utilized to display the data on toxicity reported by participants.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Stratum A: Newly Diagnosed DIPG | Stratum B: Newly Diagnosed Glioma (Non-DIPG) | Stratum C: Newly Diagnosed DIPG or Other Midline Glioma
Number analyzed (Participants) | 19 | 10 | 21
percentage of participants
  Abdominal Pain | 5.26 | 0 | 0
  Abducens Nerve Disorder | 21.0 | 0 | 9.5
  Acoustic Nerve Disorder | 5.26 | 0 | 0
  Adult respiratory distress syndrome | 0 | 0 | 4.8
  Agitation | 10.5 | 0 | 0
  Alanine aminotransferase increased | 42.1 | 20 | 28.6
  Alkalosis | 5.26 | 0 | 0
  Allergic Reaction | 0 | 10 | 4.8
  Alopecia | 0 | 0 | 9.5
  Anemia | 15.8 | 10 | 14.3
  Anorexia | 5.26 | 20 | 23.8
  Arthralgia | 15.8 | 0 | 0
  Aspartate aminotransferase increased | 36.8 | 20 | 19
  Aspiration | 5.26 | 0 | 4.8
  Ataxia | 10.5 | 0 | 0
  Atelectasis | 5.26 | 0 | 0
  Blood bicarbonate decreased | 0 | 0 | 4.8
  Blood bilirubin increased | 0 | 10 | 0
  Blurred Vision | 5.26 | 0 | 0
  Bruising | 5.26 | 0 | 0
  Cardiac troponin T increased | 0 | 0 | 9.5
  Chills | 5.26 | 0 | 0
  Constipation | 0 | 0 | 14.3
  CPK increased | 0 | 0 | 4.8
  Creatinine Increased | 5.26 | 0 | 4.8
  Depressed levels of consciousness | 5.26 | 0 | 0
  Diarrhea | 10.5 | 10 | 0
  Dizziness | 5.26 | 0 | 14.3
  Dry Skin | 0 | 0 | 4.8
  Dysarthria | 15.8 | 0 | 23.8
  Dysphagia | 10.5 | 0 | 14.3
  Dysphasia | 5.26 | 0 | 9.5
  Dyspnea | 0 | 0 | 4.8
  Edema Cerebral | 0 | 0 | 4.8
  Encephalopathy | 0 | 0 | 4.8
  Enterocolitis Infectious | 5.26 | 0 | 0
  Eosinophilia | 0 | 0 | 4.8
  Epistaxis | 5.26 | 0 | 0
  Extraocular muscle paresis | 0 | 0 | 4.8
  Eye disorders - Other | 0 | 10 | 4.8
  Facial Nerve Disorder | 5.26 | 0 | 23.8
  Fatigue | 36.8 | 50 | 61.9
  Fever | 25.3 | 30 | 28.6
  Flu like symptoms | 5.26 | 40 | 0
  Gait Disturbance | 15.8 | 10 | 4.8
  General disorders and administration site conditions - Other | 5.26 | 0 | 4.8
  Generalized Muscle Weakness | 5.26 | 0 | 4.8
  GGT Increased | 0 | 10 | 0
  Glossopharyngeal nerve disorder | 5.26 | 0 | 14.3
  Headache | 47.3 | 30 | 38
  Hearing Impaired | 0 | 0 | 4.8
  Hiccups | 5.26 | 0 | 0
  Hydrocephalus | 5.26 | 10 | 14.3
  Hyperglycemia | 5.26 | 0 | 0
  Hypernatremia | 0 | 0 | 4.8
  Hypersomnia | 5.26 | 0 | 0
  Hypertension | 0 | 0 | 14.3
  Hyperthyroidism | 0 | 0 | 4.8
  Hypoalbuminemia | 5.26 | 10 | 4.8
  Hypocalcemia | 5.26 | 10 | 0
  Hypoglycemia | 5.26 | 0 | 4.8
  Hypokalemia | 10.5 | 20 | 19
  Hypomagnesemia | 0 | 0 | 4.8
  Hyponatremia | 5.26 | 0 | 14.3
  Hypophosphatemia | 0 | 10 | 14.3
  Hypotension | 0 | 0 | 4.8
  Hypoxia | 5.26 | 10 | 0
  Injection Site Reaction | 68.4 | 50 | 38.1
  International Normalized Ratio (INR) increased | 0 | 10 | 0
  Intracranial Hemorrhage | 5.26 | 0 | 4.8
  Investigations - Other | 10.5 | 0 | 0
  Keratitis | 5.26 | 0 | 0
  Lethargy | 5.26 | 0 | 0
  Leukocytosis | 5.26 | 0 | 0
  Lipase Increased | 0 | 0 | 14.3
  Lung Infection | 10.5 | 10 | 4.8
  Lymphocyte count decreased | 31.5 | 60 | 28.6
  Lymphocyte Count Increased | 0 | 0 | 4.8
  Meningitis | 5.26 | 0 | 0
  Movements involuntary | 0 | 0 | 4.8
  Muscle Weakness Left-Sided | 21 | 0 | 19
  Muscle Weakness Right-Sided | 15.8 | 10 | 9.5
  Musculoskeletal and connective tissue disorder - Other | 5.26 | 0 | 0
  Myalgia | 15.8 | 0 | 4.8
  Myositis | 5.26 | 0 | 0
  Nasal Congestion | 5.26 | 0 | 0
  Nausea | 21 | 10 | 19
  Neck Pain | 0 | 10 | 4.8
  Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other | 0 | 20 | 4.8
  Nervous system disorders - Other | 10.5 | 0 | 23.8
  Neutrophil count decreased | 15.8 | 10 | 19
  Nystagmus | 5.26 | 0 | 9.5
  Oculomotor nerve disorder | 5.26 | 0 | 0
  Optic Nerve Disorder | 5.26 | 0 | 0
  Pain | 5.26 | 0 | 19
  Pain in extremity | 10.5 | 0 | 4.8
  Paresthesia | 5.26 | 10 | 14.3
  Platelet Count Decreased | 5.26 | 10 | 4.8
  Pruritus | 5.26 | 10 | 9.5
  Pyramidal tract syndrome | 5.26 | 0 | 0
  Rash maculo-papular | 0 | 10 | 4.8
  Renal and urinary disorders - Other | 5.26 | 0 | 0
  Respiratory failure | 0 | 0 | 4.8
  Respiratory, thoracic and mediastinal disorders - Other | 10.5 | 0 | 4.8
  Seizure | 15.8 | 0 | 0
  Skin and subcutaneous tissue disorders - Other | 10.5 | 0 | 9.5
  Skin induration | 2.63 | 10 | 14.3
  Skin Infection | 5.26 | 0 | 0
  Somnolence | 10.5 | 0 | 4.8
  Spasticity | 0 | 0 | 4.8
  Stomach Pain | 10.5 | 0 | 4.8
  Stroke | 5.26 | 0 | 0
  Thromboembolic event | 0 | 0 | 4.8
  Thyroid stimulating hormone increased | 0 | 0 | 4.8
  Trigeminal Nerve Disorder | 5.26 | 0 | 0
  Urinary Retention | 5.26 | 0 | 4.8
  Urinary Tract Infection | 5.26 | 0 | 0
  Vaccination Complication | 0 | 0 | 4.8
  Vomiting | 31.6 | 60 | 57.1
  Weight Gain | 0 | 10 | 9.5
  Weight Loss | 5.26 | 10 | 14.3
  White blood cells decreased | 31.6 | 60 | 9.5

2. Primary Outcome: Overall Survival Rate at 12 Months (OS12) (Stratum A Only)
Description: OS12 is defined as the percentage of participants still alive at 12 months, and is the clinical efficacy, primary endpoint for Stratum A. Any eligible participant that received at least one dose of the K27M/TT vaccine will be considered evaluable for clinical efficacy. OS12 will be censored at the last contact date and estimated using the Kaplan-Meier method.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum A: Newly Diagnosed DIPG
Number analyzed (Participants) | 19
percentage of participants | 42 [25 to 71]

ADVERSE EVENTS:
Time Frame: Up to 24 months
Arm/Group | Stratum A: Newly Diagnosed DIPG | Stratum B: Newly Diagnosed Glioma (Non-DIPG) | Stratum C: Newly Diagnosed DIPG or Other Midline Glioma
All-Cause Mortality (participants affected / at risk) | 17/19 | 7/10 | 20/21
Serious Adverse Events (participants affected / at risk) | 6/19 | 8/10 | 13/21
Other Adverse Events (participants affected / at risk) | 19/19 | 10/10 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A: Newly Diagnosed DIPG (N=19) | Stratum B: Newly Diagnosed Glioma (Non-DIPG) (N=10) | Stratum C: Newly Diagnosed DIPG or Other Midline Glioma (N=21)
Eye disorders - Other (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (4) | 3 (3)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness left-sided (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness right-sided (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) | 0 (0) | 5 (5)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A: Newly Diagnosed DIPG (N=19) | Stratum B: Newly Diagnosed Glioma (Non-DIPG) (N=10) | Stratum C: Newly Diagnosed DIPG or Other Midline Glioma (N=21)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 2 (10) | 4 (7)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Hearing Impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 1 (2) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other (Eye disorders) | 2 (2) | 1 (2) | 2 (3)
Eye Pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Flashing lights (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 2 (3) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Papilledema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 5 (8)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (4) | 0 (0) | 2 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (10) | 1 (1) | 6 (10)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (14) | 6 (10) | 11 (15)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 10 (10) | 5 (10) | 14 (25)
Fever (General disorders) | 6 (10) | 3 (4) | 6 (7)
Flu like symptoms (General disorders) | 1 (1) | 4 (7) | 0 (0)
Gait disturbance (General disorders) | 5 (6) | 3 (3) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 13 (24) | 5 (6) | 8 (10)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (2) | 0 (0) | 4 (4)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (3) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 8 (14) | 4 (5) | 7 (15)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 8 (12) | 2 (2) | 4 (10)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Blood bilirubin increased (Investigations) | 1 (3) | 1 (2) | 0 (0)
Cardiac troponin T increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 1 (1)
CPK increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 1 (1) | 1 (3)
Fibrinogen decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other (Investigations) | 2 (55) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 3 (4)
Lymphocyte count decreased (Investigations) | 7 (16) | 6 (18) | 11 (21)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3) | 1 (1) | 4 (8)
Platelet count decreased (Investigations) | 1 (2) | 1 (9) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 2 (2) | 5 (8)
Weight loss (Investigations) | 3 (4) | 2 (2) | 4 (8)
White blood cell decreased (Investigations) | 6 (9) | 7 (13) | 6 (11)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (6) | 1 (1) | 3 (5)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 2 (3)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (10) | 1 (2) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 5 (7) | 2 (3) | 5 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 3 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 4 (7)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle weakness left-sided (Nervous system disorders) | 5 (6) | 0 (0) | 4 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness right-sided (Nervous system disorders) | 3 (3) | 0 (0) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 1 (3)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 6 (7) | 2 (2) | 7 (10)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 6 (7)
Dysarthria (Nervous system disorders) | 3 (3) | 0 (0) | 6 (9)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 3 (4)
Edema cerebral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 3 (3) | 1 (2) | 6 (8)
Glossopharyngeal nerve disorder (Nervous system disorders) | 1 (4) | 1 (1) | 4 (5)
Headache (Nervous system disorders) | 11 (14) | 4 (7) | 8 (26)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
IVth nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 2 (5) | 2 (2) | 1 (1)
Nystagmus (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Oculomotor nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 1 (3) | 3 (4)
Pyramidal tract syndrome (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Glucosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (3)
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (3) | 1 (1) | 1 (2)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 2 (3)
Skin induration (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (2) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (3) | 4 (4) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT02960230/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT02960230/ICF_001.pdf